CLINICAL TRIAL: NCT06529094
Title: Implementing a Decision Support Tool to Prevent Community-Acquired Pressure Injury in Spinal Cord Injury (SCI) in the Spinal Cord Injury Clinic
Acronym: CAPP-FIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); VA Long Beach Healthcare System (U.S. Federal Agency); Saint Louis VA Medical Center (U.S. Federal Agency); James A. Haley Veterans' Hospital (Unknown); Louis Stokes VA Medical Center (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Iowa City Veterans Affairs Medical Center (U.S. Federal Agency); San Diego Veterans Healthcare System (U.S. Federal Agency); Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IIR 22-163; HX003704 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2024-07-16; First posted 2024-07-31 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury; Pressure Injury
Keywords: prevention; spinal cord injury; pressure injury; Veteran; community
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The RE-AIM (Reach, Efficacy, Adoption, Implementation, and Maintenance) framework will guide this study to assess implementation. For this study, Reach is the proportion of the outpatient SCI population that complete the CAPP-FIT. Efficacy is success rate, measured as reduction in incidence of CAPrIs, CAPrI-associated hospitalizations, and patient and provider satisfaction. Adoption is the degree that sites use the CAPP-FIT. Implementation is the extent to which the CAPP-FIT is implemented as intended. Maintenance is the extent to which CAPP-FIT is maintained over time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Preparation to implement the CAPP-FIT per site (Other): Complete clinic workflow designs and redesigns to integrate CAPP-FIT into clinic workflow per site. Recruit and train providers in use of the CAPP-FIT through TMS training, demonstration, and simulation with a standardized patient.
  Interventions: Behavioral: Provider training
- Implement CAPP-FIT with RA facilitation (Active Comparator): Veteran completes Veteran Survey and Provider uses Provider report around an established clinic visit per site
  Interventions: Behavioral: CAPP-FIT intervention with RA facilitation
- Implement CAPP-FIT without RA facilitation (Other): Each site will determine how they will integrate use of the CAPP-FIT in clinic workflow.
  Interventions: Behavioral: CAPP-FIT implementation during maintenance phase

INTERVENTIONS:
Behavioral: Provider training — Provider participants will complete TMS training, CAPP-FIT demonstration and simulation in use of the CAPP-FIT with a standardized patient.
  Arms: Preparation to implement the CAPP-FIT per site
Behavioral: CAPP-FIT intervention with RA facilitation — After consent and survey completion, RA to email/text CAPP-FIT link to Veteran the day before established clinic visit. RA to remain available to answer questions to help Veteran participant complete Veteran Survey and submit the responses through eScreening. The Provider Report will appear in CPRS with a Provider notification. RA to meet Veteran participant in the clinic after the clinic visit to complete the Veteran satisfaction survey.
  Arms: Implement CAPP-FIT with RA facilitation
Behavioral: CAPP-FIT implementation during maintenance phase — Providers will attend focus group after Arm 2 to determine sustainability of CAPP-FIT use in clinic workflow. Clinic provider will act on that determination for 10 months during maintenance phase.
  Arms: Implement CAPP-FIT without RA facilitation

SUMMARY:
Spinal cord injury (SCI) is a permanent condition affecting every aspect of life including health, daily activities, and participation and quality of life. Persons with SCI are at high risk of pressure injury (PrI) throughout their lives due to loss of sensation, nerve damage and immobility. PrIs are local areas of damage to the skin and underlying soft tissue caused by pressure and shear commonly located over bony prominences. While most PrIs are hospital- or nursing home-acquired, in people with SCI, PrIs typically develop in the community. Community-acquired pressure injuries (CAPrIs) are common, devastating, and costly. This grant proposal will assess how well a decision support tool, called the Community Acquired Pressure Injury Prevention Field Implementation Tool (CAPP-FIT), is used in the clinic and how well it prevents CAPrIs. The CAPP-FIT will be implemented at seven sites across the country in a staggered fashion. The CAPP-FIT includes: 1) an automated Veteran survey to identify risks, actions, and resources needed to prevent CAPrIs and 2) a companion Provider Report immediately available in the electronic health record listing Veteran responses to survey items with recommended evidence-based provider actions. The Veteran survey can be completed via a secured email on the computer or phone. There are three aims in the proposal: Aim 1 is implementing the CAPP-FIT at the seven geographically diverse VA SCI clinics. After CAPP-FIT implementation, each site will determine how the CAPP-FIT will be maintained in clinical practice to support sustainability. Aim 2 assesses how well the CAPP-FIT prevents CAPrIs and CAPrI-associated hospitalizations and assesses provider and Veteran satisfaction. Aim 3 assesses how well the CAPP-FIT is implemented in the SCI clinic.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a permanent condition affecting every aspect of life including health, daily activities, and participation and quality of life. Persons with SCI are at high risk of pressure injury (PrI) throughout their lives due to loss of sensation, nerve damage and immobility. PrIs are local areas of damage to the skin and underlying soft tissue caused by pressure and shear commonly located over bony prominences. While most PrIs are hospital- or nursing home-acquired, in people with SCI, PrIs typically develop in the community. Community-acquired pressure injuries (CAPrIs) are common, devastating, and costly. This grant proposal is a type 1 hybrid stepped wedge randomized design at six additional SCI Clinics to assess the efficacy and implementation of a decision support tool, called the Community Acquired Pressure Injury Prevention Field Implementation Tool (CAPP-FIT) previously developed and piloted at one site. The CAPP-FIT includes: 1) a Veteran survey to identify risks, actions, and resources needed to prevent CAPrIs and 2) a companion Provider Report immediately available in print or downloaded into the electronic health record listing Veteran responses to survey items with recommended evidence-based provider actions. The Veteran survey can be completed at home via a secured email or by using an iPad in the clinic. There are three aims in the proposal, guided by the RE-AIM framework. Aim 1 is implementing the CAPP-FIT at the seven geographically diverse VA SCI clinics, including workflow redesign, provider training, and evaluation of provider readiness. The CAPP-FIT will be implemented in a staggered fashion consistent with the stepped wedge design. After CAPP-FIT implementation, each site will determine how the CAPP-FIT will be maintained in clinical practice to support sustainability (maintenance phase). Aim 2 assesses efficacy, assessing provider and Veteran satisfaction in CAPrI use, new CAPrI incidence for 6 months post-initial CAPP-FIT implementation, and overall and CAPrI-associated hospitalizations. Aim 3 assesses implementation using RE-AIM. Reach is the proportion of providers and Veterans participating in the intervention. Adoption is assessed by the proportion of Veteran-identified modifiable risk factors acted upon by SCI providers, as well as a comparison of non-modifiable risk factors of participating and non-participating VA SCI clinics. Implementation is assessed by describing completed CAPP-FITs during implementation, describing Veteran CAPrI risk factors, and describing provider identified facilitators and barriers to implementation. Maintenance is assessed by describing how each clinic will continue to integrate CAPP-FIT into workflow and by describing the number of providers using the CAPP-FIT during maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

Veteran participant eligibility criteria include:

* assigned provider in SCI clinic who is willing to participate in the study
* has a scheduled appointment in the SCI clinic
* ability to complete survey

Exclusion Criteria:

* active diagnosis of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of new community acquired pressure injury 6 months post CAPP-FIT implementation | 6 months
  New CAPrI incidence within 6 months of first CAPP-FIT survey measured for each unique patient

SECONDARY OUTCOMES:
Root causes of new CAPrIs that occur 6 months post CAPP-FIT implementation | 6 months
  Use of root cause analysis (RCA) to determine the cause of a new CAPrIs within 6 months post CAPP-FIT implementation in Veteran participants
Veteran satisfaction with the CAPP-FIT Information | after first CAPP-FIT completion-month 5 through 35
  Veteran satisfaction with the initial use of the CAPP-FIT will be assessed using the Information subscale of the Mobile Application Rating Scale (MARS), which rates the six items of a 5-point scale from 1 (inadequate) to 5 (excellent). Minimum score is 6, maximum score is 30.
Provider satisfaction with CAPP-FIT | Month 35-36 and month 45-46 (after implementation and after maintenance phases)
  The investigators will hold focus groups with providers per site after implementation to evaluate provider satisfaction with the CAPP-FIT. The investigators anticipate focus groups to include approximately 6-12 participating interprofessional providers/site. Each focus group will be audiotaped and transcribed verbatim. Data will be analyzed using content analysis to identify themes that emerge from the data per site. Qualitative coders will independently code the focus group data, meet to discuss codes, and discrepancies and come to consensus to develop the codebook and finalize themes.
Inpatient admissions and PrI-associated inpatient admissions | 6 months post initial CAPP-FIT implementation
  The incidence of inpatient admission within 6 months of first CAPP-FIT survey measured for each unique patient over time. Covariates of interest include non-modifiable CAPrI risk factors.
Proportion of SCI providers that attend training and simulation | prior to CAPP-FIT implementation
  The investigators will obtain a roster of all providers who see patients in the SCI clinic (denominator). Those who agree to participate in the study will be the numerator to determine reach, such that the proportion of the target population participating in the intervention is calculated as the numerator divided by the denominator.
Proportion of Veteran participants completing CAPP-FIT during study periods | after Veteran CAPP-FIT completion (Months 5 through 35)
  The number of unique patients that meet inclusion criteria and have completed clinic appointments with participating providers during data collection periods is the denominator. Those who agree to participate in the study and complete the CAPP-FIT eScreening will be the numerator. Veteran reach is calculated as the numerator divided by the denominator.
Veteran risk factors identified per site during CAPP-FIT implementation | after Veteran CAPP-FIT completion (Months 5 through 35)
  Veteran identified risk factors will be collected from the Provider Report in RedCap. Risk factor categories are issues associated with pressure reduction, nutrition, access to care, skincare, incontinence, acute illness, coping/motivation, mobility/activity, repositioning, caregiver, life integration, and substance use.
Provider actions on Veteran risks identified on the Veteran survey during implementation | One week after Veteran CAPP-FIT completion/Provider Report generation (month 5 through 36)
  Chart review will reveal whether recommended provider actions listed on the Provider Report for Veteran-identified risk factors were addressed at or within one week of CAPP-FIT completion during a clinic visit.
Completed Veteran survey and accessed Provider Reports during implementation | Day of CAPP-FIT completion (month 5-35)
  Proportion of completed Veteran surveys that Providers accessed during implementation.
Describe and compare the patient population of participating VA SCI Centers: Healthcare access (travel time) | 6 months after CAPP-FIT completion (month 5-35)
  Description and comparison of Veterans who have an assigned primary care provider in the SCI Clinic on non-modifiable characteristics that affect CAPrI incidence: healthcare access (travel time). Travel time from home to nearest VA Hospital.
Facilitators/barriers in implementing the CAPP-FIT per site | monthly to 6-weeks (month 5-35), at end of implementation (month 35-36) and maintenance phases (Month 45-46)
  Contextual inquiry will be conducted four times a month per site during implementation to identify identify implementation barriers including fidelity in CAPP-FIT use. Contextual summaries will be shared and discussed with providers during each site provider group monthly to 6 week meetings and discuss facilitators, barriers, and possible recommended changes to workflow, patient flow in implementation. Meeting minutes will be maintained. A focus group of provider participants per site will be conducted at the end of implementation and maintenance to evaluate provider satisfaction, facilitators, and barriers to implement the CAPP-FIT. Focus groups will be audiotaped, transcribed, and verified and analyzed by two qualitative researchers.
Description of how sites will maintain the CAPP-FIT in clinic workflow post implementation | end of implementation (month 35-36) and maintenance phases (months 45-46)
  The end-of-implementation provider focus group will reveal how the CAPP-FIT will be maintained in clinic workflow. This includes any change in adapting the CAPP-FIT to clinic practice, changed workflow, and implementation protocols. This assessment will be repeated during the end-of-maintenance focus group.
Describe and compare the patient population of participating VA SCI Centers: Medium and Dark Skin Tone | At initial CAPP-FIT completion (month 5-35)
  Description and comparison of Veterans who have an assigned primary care provider in the SCI Clinic on non-modifiable characteristics that affect CAPrI incidence: African-American/non-African-American
Describe and compare the patient population of participating VA SCI Centers: Level of Injury | at initial CAPP-FIT completion (month 5-35)
  Description and comparison of Veterans who have an assigned primary care provider in the SCI Clinic on non-modifiable characteristics that affect CAPrI incidence: tetraplegia or paraplegia
Describe and compare the patient population of participating VA SCI Centers: history of pressure injury | At initial CAPP-FIT completion (month 5-35)
  Description and comparison of Veterans who have an assigned primary care provider in the SCI Clinic on non-modifiable characteristics that affect CAPrI incidence: a documented pressure injury within 5 years prior to the initial CAPP-FIT completion.
Describe and compare the patient population of participating VA SCI Centers: Age | at initial CAPP-FIT completion (month 5-35)
  Description and comparison of Veterans who have an assigned primary care provider in the SCI Clinic on non-modifiable characteristics that affect CAPrI incidence: age in years
Describe and compare the patient population of participating VA SCI Centers: Care Assessment Needs (CAN score) | At initial CAPP-FIT completion (month 5-35)
  Description and comparison of Veterans who have an assigned primary care provider in the SCI Clinic on non-modifiable characteristics that affect CAPrI incidence: CAN score. CAN score is risk of hospitalization in 90 days. The score also compares the Veteran with other individuals and ranks them in a percentile from zero (lowest risk) to 99 (highest risk).
Describe and compare the patient population of participating VA SCI Centers: ASIA Impairment Scale score | At initial CAPP-FIT completion
  Description and comparison of Veterans who have an assigned primary care provider in the SCI Clinic on non-modifiable characteristics that affect CAPrI incidence: ASIA Impairment Scale (AIS) measures functional impairment due to the spinal cord injury. Grade A=The impairment is complete. There is no motor or sensory function left below the level of injury. Grade B=The impairment is incomplete. Sensory function, but not motor function, is preserved below the neurologic level and some sensation is preserved in the sacral segments S4 and S5. Grade C=Motor function is preserved below the neurologic level and not strong enough to move against gravity. Grade D: The impairment is incomplete. Joints can move against gravity. Grade E: functions are normal.
Veteran satisfaction with the CAPP-FIT Functionality | after first CAPP-FIT completion-month 5 through 35
  Veteran satisfaction with the initial use of the CAPP-FIT will be assessed using the Functionality subscale of the Mobile Application Rating Scale (MARS), which rates the five items of a 5-point scale from 1 (inadequate) to 5 (excellent). Minimum score is 5, maximum score is 25.
Veteran Satisfaction with healthcare | immediately prior to first CAPP-FIT completion (month 5 through 35) and six months after first CAPP-FIT completion (month 11 - 41)Implemen and again at the end of
  Veteran satisfaction with healthcare will be measured pre and 6 months post CAPP-FIT intervention using the Scale of Patient Satisfaction with Primary Care Provider, which is a 10-item scale measured on 7-point Likert scale (1=strongly disagree, 7=strongly agree). Minimum value is 7; maximum value is 70.
Change in proportion of NP/MD/RN providers implementing the CAPP-FIT between implementation and maintenance | end of implementation months (month 5-35) and maintenance phases (month 36-45)
  The number of providers per site who access the CAPP-FIT during implementation and maintenance phases (numerator). Total number of providers at each site (denominator). The comparison is the change in proportion of providers who use the CAPP-FIT at each site.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Burkhart, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (7):
- United States (7):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the proposed research will be shared outside VA.
  A de-identified, anonymized dataset will be created and shared. The VA privacy officer will certify whether the data sets meet conditions for disclosure to the public within one year of publication. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by ORD. Those requesting data will be asked to sign a Data Use Agreement (DUA) in compliance with VA and non-VA privacy regulations.
  Documentation will accompany each dataset. The analytical datasets and statistical code used in the publication will be retained for 6 years, in accordance with VA record retention policy.
Supporting Information: Study Protocol, SAP
Time Frame: The analytical datasets and statistical code used in the publication will be retained for 6 years, in accordance with VA record retention policy.
Access Criteria: Data will become available at the end of the study. The analytical datasets and statistical code used in the publication will be retained for 6 years, in accordance with VA record retention policy.